CLINICAL TRIAL: NCT03501433
Title: Effects of Nicotinamide Riboside on Metabolism and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Rudy Valentine, Assistant Professor, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-603
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Aging; Lipemia
Keywords: postpandial; lipemia; microvascular
MeSH Terms: conditions — Hyperlipidemias | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over
Who Masked: Participant, Outcomes Assessor
Masking Description: I single investigator will be responsible for blinding. All researchers involved in collection and evaluation of data will remain blinded to treatments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide Riboside Chloride (Niagen) (Experimental): 7 days of nicotinamide riboside supplementation (250 mg/d x 2/day).
  Interventions: Dietary Supplement: Nicotinamide riboside chloride (Niagen)
- Placebo (Placebo Comparator): 7 days of placebo supplementation (2/day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide riboside chloride (Niagen) — 250 mg capsules 2x/day for 7 days
  Other Names: Nicotinamide Riboside, Niagen
  Arms: Nicotinamide Riboside Chloride (Niagen)
Dietary Supplement: Placebo — 2x/day for 7 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of Nicotinamide Riboside (NR) supplementation on metabolism and vascular function following high-fat meal. Differences between young (18-35) and older (60-75) adults will be determined.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of 7 days of Nicotinamide Riboside (NR) or placebo supplementation on metabolism and vascular function following high-fat meal. Differences between young (18-35) and older (60-75) adults will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35 (young) and 60 to 75 (older)
* Normo- or pre-hypertensive (blood pressure <140/90 mmHg)
* Non-smokers
* Able to give informed consent and participate in all laboratory visits

Exclusion Criteria:

* Currently taking any medications that could interfere with cardiovascular or metabolic outcomes will be excluded from the study (e.g., beta-blockers)
* Known metabolic (e.g. Type I or Type II diabetes, cardiovascular disease, etc.) or immunologic (e.g. HIV, cancer, autoimmune, etc.) diseases
* Food allergies to egg, milk, soy or wheat
* Women who are pregnant or planning to become pregnant during the course of the study,
* Pacemaker or other implanted device
* Unwilling to participate in the experimental protocol or blood draws will be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
NAD+ | 7 days
  Blood and peripheral blood mononuclear cell (PBMC) levels

SECONDARY OUTCOMES:
Vasodilatory responsiveness | 7 days
  Post-Occlusion Reactive Hyperemia (PORH)
Lipdemia | 7 days
  Fasting and postprandial
Oxidative stress and inflammation | 7 days
  Plasma markers and expression in circulating PBMCs

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Valentine, PhD, Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: No